CLINICAL TRIAL: NCT04746599
Title: Autologous Fat Grafting in the Treatment of Critical Limb Ischaemia Non Suitable for Revascularization: The Adipose Tissue - Critical Limb Ischaemia (ADIPOCLI) Trial Protocol
Brief Title: Autologous Fat Grafting in the Treatment of Critical Limb Ischaemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1130
Record Dates: First submitted 2021-02-03; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Critical Limb Ischemia; Peripheral Arterial Disease - PAD; Ischemic Ulcer; Ischemic Feet; Diabetic Foot; Scleroderma, Systemic; Thrombo Angiitis Obliterans; Ischemic Leg
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Diabetic Foot; Scleroderma, Systemic; Thromboangiitis Obliterans

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with critic limb ischemia (Experimental): Patient enrolled from emergency room or outpatient population undergo pre-operatory tests including blood test, thoracic radiography, electrocardiogram, cardiologic visit, TcPO2 measurement and Doppler ultrasonography. During surgery the terminal branches of the patient's leg arteries are mapped and under local anesthesia multiple injections (1 mL each) of the adipose tissue formulation are inoculated 1 cm above the end of the terminal branch of the peroneal, anterior, and posterior tibial arteries. Furthermore, a total amount of 0.5-1 ml of the autologous adipose tissue-derived cell (ATDC) fraction is injected 1 cm near to ischaemic lesions.
  After the surgical procedure, the patient will be followed for 6 months, during which he will undergo outpatient visits at 7 and 21 days; then at 1, 3 and 6 months. At each visit, the patient will be assessed for the amount of pain, the transcutaneous oximetry value, measurement of the ABI index, arterial ultrasound Doppler lower limbs.
  Interventions: Procedure: Autologous Fat Grafting

INTERVENTIONS:
Procedure: Autologous Fat Grafting — The trochanteric area or the periumbilical abdominal region represents the donor sites. Following Coleman's technique and after the administration of modified Klein solution, a skin incision is performed in the selected area. Adipose tissue is harvested and after suture the area is managed with an elastic-compressive dressing, to be kept in place for 5 days to prevent hematoma formation. The adipose tissue is the centrifuged at 920 × g for 3 min in sterile conditions. Only the intermediate layer containing adipocytes and stromal vascular component will be then injected using a blunt cannula. The terminal branches of the patient's leg arteries are mapped to facilitate graft placement. Under local anesthesia multiple injections of the adipose tissue formulation are inoculated 1 cm above the end of the terminal branch of the peroneal, anterior, and posterior tibial arteries.
  Other Names: adipose tissue transplantation

SUMMARY:
Critical Limb Ischaemia (CLI) is a condition characterized by chronic ischemic at-rest pain, ulcers, or gangrene for more than 2 weeks in one or both legs, attributable to objectively proven arterial occlusive disease.CLI is associated with a high risk of lower amputation, diminished quality of life and mortality. Revascularization by either bypass surgery or endovascular recanalization is considered the first-choice treatment in patients with CLI.

Revascularization is not always possible because patients with CLI often have severe comorbidities or because it is not technically feasible.

On the basis of their well-recognized regenerative and angiogenetic properties, cell therapy with autologous bone marrow-derived mesenchymal stem cells (BMMSCs) has been proposed and tested in different animal models and in some human pathological conditions characterized by peripheral ischemia and wound formation.

DETAILED DESCRIPTION:
The ADIPOCLI trial is an interventional monocentric trial in which the investigators will evaluate the safety, feasibility and potential efficacy of local administration of autologous adipose derived stromal/stem (ASCs) cell as treatment for pain and ulcers caused by CLI. If the results confirm safety, feasibility and show potential beneficial effects of the intervention regarding clinical parameters, a larger clinical research with longer follow up will be initiated focusing on efficacy. The objective of this clinical trial is to assess the efficacy and safety of ASCs inoculation in peri-tibial area, though reducing pain significantly in patients with CLI not eligible for revascularization.

Autologous fat grafting is widely used for soft-tissue augmentation and replacement in reconstructive and aesthetic surgery providing a biocompatible, natural and inexpensive method. Noteworthy, recent reports have identified adipose tissue as the tissue in the body that contains the highest percentage of adult stem cells. These adipose derived stem cells (ADSCs) can undergo multilineage differentiation and may be crucial for the surgery purpose of healing ulcers as they have potent regenerative effects on endothelium and immunomodulatory properties.

Adipose-derived stromal/stem cells (ASCs) are considered to be an attractive alternative to pluripotent cells with characteristics similar to BMMSCs. Compared with these latter cells, ASCs offer several advantages, including ease of isolation, less donor morbidity, relative abundance, and rapidity of expansion. Preliminary attempts with ASC cell therapy have been made to induce healing of ulcers developed in peripheral vascular diseases of some animal models and human disorders.

The benefits of peritibial inoculation of autologous adipose tissue are the reduction of ischemic pain, the improvement of skin and muscle perfusion, the suspension of major amputation interventions and the healing of trophic lesions if present.

The result of the intervention varies from individual to individual and depends on the engraftment of the transplanted material. In some cases the pain completely disappears. In others, the transplanted material may undergo varying degrees of reabsorption (from 50% to 70%) and therefore a new transplant may be necessary after some time (6-12 months).

The risks are linked to local complications of the procedure such as edema, ecchymosis, pain in the district of surgical aggression (the extent of these three manifestations varies from patient to patient, but are generally modest), dehiscence, bleeding of the wound, site infection surgical.

The study has a total duration of 24 months. The recruitment phase lasts 18 months. After the surgical procedure, the patient will be followed for 6 months, during which he will undergo outpatient visits at 7 and 21 days; then at 1, 3, and 6 months. At each visit, the patient will be assessed for the amount of pain and the transcutaneous oximetry value. As in the usual clinical practice and in the diagnostic-therapeutic path of the arteriopathic patient, instrumental examinations (measurement of the ankle-brachial pressure index - ABI, arterial ultrasound Doppler lower limbs) are performed at the enrollment, at the twenty-first day and 6 months after the procedure .

The investigators will include 20 patients with CLI who satisfy the inclusion criteria. Inclusion and exclusion criteria were designed to select patients with CLI, not suitable for revascularization and who are in reasonable health condition to allow trial participation. Study participants are recruited from our own outpatient population or emergency room. Baseline characteristics are collected during the first visit and include medical examination, ABI and TcPO2 evaluation and Doppler ultrasonography to study the arterial axis of the limb. If CLI is diagnosed, the patient is hospitalized and undergoes an angiography study. Quality of Lyfe test is administered at hospitalization and at follow up.

After angiogram, treatment of choice will be selected during the multidisciplinary vascular conference taking the individual condition of patients into account. Patients eligible for revascularization are submitted to open/endovascular surgery. Patient with CLI unsuitable for revascularization continue hospitalization being given best medical therapy, i.e. pain-killer drugs and prostanoids. Only to these class of patients an adjunctive treatment with local fat grafting is proposed. Information sheet is given to every patient after interview with investigators and informed consent is taken before the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Established diagnosis of CLI according to TransAtlantic InterSociety Consensus (TASC II) guidelines
* Ankle oxygen partial pressure < 40 mmHg with no ischaemic lesions or < 60 mmHg with ischaemic lesions
* Tibial injections site free from ulcers
* Absence of comorbidities responsible for life expectancy < 6 months
* Non suitability for surgery (comorbidities or angiographic results)
* Informed consent taken

Exclusion Criteria:

* Age < 18 years
* Inability of understanding and signing informed consent
* Tibial injections sites involved by ulcers
* Life expectancy < 6 months
* Unwillingness to attend follow up
* Any of the following: women who are or may be pregnant or women hoping to become pregnant; women who are breastfeeding; men whose partners hope to become pregnant during the treatment period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain reduction | 7 days
  Primary endpoint is pain change or complete disappearance, according to Numeric Rating Scale (NRS) ranging from 0 (no pain) ad 10 (maximum amount of pain), ad TcPO2 improvement. The investigators will consider significative a pain change below NRS<4 and a improvement in TcPO2 (> 40 mmHg in patients with rest pain and no ischaemic lesions or > 60 mmHg in patients with rest pain and ischaemic lesions) among at least 70% (14) of the patients enrolled in the study.

SECONDARY OUTCOMES:
Limb salvage | 30 days
  Secondary endpoint is a change in limb salvage rate > 50%, compared to Literature. Literature suggests that a year after the onset of CLI, only about half the patients will be alive without a major amputation, although some of these may still have rest pain, gangrene or ulcers. Approximately 25% will have died and 25% will have required a major amputation. Again, in contrast to patient with intermittent claudication, patients with CLI are on a rapidly downward course in term of both life and their prognosis is in many ways similar to that of some malignant forms of cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Santi Trimarchi, Prof, Principal Investigator — Fondazione IRCCS Cà Granda Ospedale Maggiore
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore di Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No